CLINICAL TRIAL: NCT06982118
Title: Investigation of the Relationship Between the Frequency of Lumbar Facet Tropism and Disc Herniation and Spondylolisthesis in Patients With Low Back Pain Complaints
Brief Title: Facet Tropism in Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, MD, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPRMTRH-EK3
Record Dates: First submitted 2025-05-08; First posted 2025-05-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain; Spondylolisthesis; Degenerative Disc Disease, Lumbar
Keywords: facet tropism; low back pain; physical therapy; magnetic resonance imaging
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with low back pain: Between 01/11/2023-01/05/2025, patients who applied to Istanbul Physical Therapy and Rehabilitation EAH Physical Medicine and Rehabilitation outpatient clinic with the complaint of low back pain and outpatient clinic archive files will be included in the study in accordance with the inclusion and exclusion criteria. Demographic data (age, gender), etiopathology (lumbar disc herniation, spondylosis, spondylolisthesis etc.), physical therapy modalities and drug use information will be noted from the archive files. The presence/grade of disc herniation, presence of spondylolisthesis and facet measurements of lumbar MRI patients registered in the hospital imaging system will be recorded. The data will be statistically analyzed and the relationship between facet tropism, disc herniation and listhesis will be tested.

SUMMARY:
This retrospective study investigates the relationship between lumbar facet tropism and the occurrence of disc herniation and spondylolisthesis in patients with low back pain who underwent lumbar MRI. Facet tropism, defined as asymmetrical facet joint rotation, is hypothesized to influence spinal biomechanics and contribute to degenerative processes. The study will evaluate MRI scans of patients with low back pain to determine the presence of facet tropism, disc herniation, and listhesis at L3-L4, L4-L5, and L5-S1 levels, aiming to identify potential associations between these conditions at various spinal levels.

DETAILED DESCRIPTION:
Background: Lumbar facet tropism refers to an asymmetry in the orientation of the facet joints within the axial plane of the lumbar spine. It is theorized that this anatomical variation can alter the biomechanics of the spine, potentially predisposing it to degenerative changes.

The literature suggests a possible association between facet tropism and lumbar disc pathologies, especially disc herniation and degeneration. Furthermore, asymmetry in the facet joints has been proposed as a factor that might contribute to the development of spondylolisthesis, defined as the forward slippage of one vertebra over another. This instability in the spine can lead to low back pain and other related clinical symptoms. However, the precise nature and strength of the relationship between facet tropism and these degenerative spinal conditions remain unclear.

To address this, the current retrospective study will examine patients who presented to a Physical Medicine and Rehabilitation outpatient clinic reporting low back pain and who subsequently underwent lumbar Magnetic Resonance Imaging (MRI). The MRI images of these patients will be analyzed to identify the presence of facet tropism, disc herniation, and spondylolisthesis at the L3-L4, L4-L5, and L5-S1 spinal levels.

This retrospective study aims to explore the potential link between lumbar facet tropism and the presence of both lumbar disc herniation and spondylolisthesis in individuals experiencing low back pain.

Methods:Between 01/11/2023-01/05/2025, patients who applied to Istanbul Physical Therapy and Rehabilitation Training and Research Hospital Physical Medicine and Rehabilitation outpatient clinic with the complaint of low back pain and outpatient clinic archive files will be included in the study in accordance with the inclusion and exclusion criteria. Demographic data (age, gender), etiopathology (lumbar disc herniation, spondylosis, spondylolisthesis etc.), physical therapy modalities and drug use information will be noted from the archive files. The presence/grade of disc herniation, presence of spondylolisthesis and facet measurements of lumbar MRI patients registered in the hospital imaging system will be recorded. The data will be statistically analyzed and the relationship between facet tropism, disc herniation and listhesis will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-80 years
* Patients admitted to the outpatient clinic with complaints of low back pain
* Patients with complete demographic and clinical data in their archive files
* Patients with lumbar MRI registered in the hospital imaging system after clinic admission

Exclusion Criteria:

* Patients with a history of lumbar surgery
* History of trauma in the lumbar region
* Active inflammatory joint disease
* Patients with central nervous system diseases such as Parkinson's disease, multiple sclerosis
* Malignancy
* Files with missing archive file records

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the physical medicine and rehabilitation outpatient clinic of Istanbul Physical Therapy and Rehabilitation Training and Research Hospital with the complaint of low back pain between 01/11/2023-01/05/2025
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of Facet Tropism | Baseline
  The presence of facet tropism at the L3-L4, L4-L5 and L5-S1 levels will be determined in patients who present with low back pain and have lumbar magnetic resonance imaging.

SECONDARY OUTCOMES:
Frequency of Lumbar Disc Herniation and Spondylolisthesis | Baseline
  The presence of disc herniation and listhesis at the L3-L4, L4-L5 and L5-S1 levels will be determined in patients who present with low back pain and have lumbar magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Therapy Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data supporting the findings of this study are available from the corresponding author upon reasonable request. However, due to patient confidentiality and ethical restrictions, the data are not publicly available.

REFERENCES:
- [Background] Kong MH, He W, Tsai YD, Chen NF, Keorochana G, Do DH, Wang JC. Relationship of facet tropism with degeneration and stability of functional spinal unit. Yonsei Med J. 2009 Oct 31;50(5):624-9. doi: 10.3349/ymj.2009.50.5.624. Epub 2009 Oct 20. PMID 19881964
- [Background] Garg K, Aggarwal A. Facet Tropism in Lumbar Spine and Cervical Spine: A Systematic Review and Meta-Analysis. World Neurosurg. 2021 Mar;147:47-65. doi: 10.1016/j.wneu.2020.11.171. Epub 2020 Dec 9. PMID 33309642
- [Background] Do DH, Taghavi CE, Fong W, Kong MH, Morishita Y, Wang JC. The relationship between degree of facet tropism and amount of dynamic disc bulge in lumbar spine of patients symptomatic for low back pain. Eur Spine J. 2011 Jan;20(1):71-8. doi: 10.1007/s00586-010-1558-8. Epub 2010 Aug 25. PMID 20734211